CLINICAL TRIAL: NCT00701272
Title: FGL2/Fibroleukin and Hepatitis C Virus Infection: A Predictor of HCV Recurrence and Progression Post Liver Transplantation
Brief Title: FGL2/Fibroleukin and Hepatitis C Virus Recurrence Post Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 08-0385-T
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Liver Transplantation; Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples; liver biopsy tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients undergoing liver transplant for end-stage liver disease due to Hepatitis C
- 2: Control population:
  Patients undergoing liver transplantation for end-stage liver disease due to alcoholic cirrhosis

SUMMARY:
The main objective of this study is to assess whether a recently-developed bioassay for the molecule "secreted fibrinogen-like protein 2" (sFGL2) can be used to predict the recurrence and/or progression of Hepatitis C Virus disease in post liver transplant patients. The hypothesis is that patients with chronic HCV have higher than normal levels of sFGL2 in their blood both pre- and post-transplantation and that this will inhibit their ability to clear HCV, and influence the progression of HCV disease when it recurs.

DETAILED DESCRIPTION:
Hepatitis C Virus infection (HCV) is a serious health problem worldwide, accounting for significant morbidity and mortality. The current treatment, combination therapy with pegylated IFNa/ribavirin results in only a 50% sustained viral response such that HCV is now the leading indication for liver transplantation. Unfortunately, HCV recurrence post-transplantation is universal and it is often difficult to distinguish recurrent HCV from other processes such as rejection, leading to inappropriate or delayed treatment(s) and compounding graft damage. It would be beneficial to have access to a circulating biomarker to distinguish HCV disease recurrence from other processes and to predict the severity of HCV disease progression post-transplantation.

The molecule FGL2 is secreted by cells of the immune system and may be a key immunomodulator affecting graft survival and HCV recurrence. The aim of this study is to assess whether a bioassay for FGL2 can predict HCV disease recurrence and progression after liver transplantation and/or differentiate HCV disease recurrence from acute cellular rejection.

This study will also examine the form of Fc Receptor expressed in these patients. The Fc receptor is hypothesized to be the binding partner of FGL2.

ELIGIBILITY:
For HCV positive subjects:

Inclusion Criteria:

1. Able and willing to give written informed consent
2. Willing to follow the study protocol
3. Diagnosis of chronic HCV infection based on two positive serology tests
4. No history of active alcohol or drug abuse
5. All six viral genotypes are considered
6. Pre- and post transplant viral load data must be available

Exclusion Criteria:

1. Pregnancy
2. HBV, HDV or HIV co-infection

For Non-HCV subjects:

Inclusion Criteria:

1. Able and willing to give written informed consent
2. Willing to follow the study protocol

Exclusion Criteria:

1. Free from infection by any of the following: HCV, HBV, HDV or HIV.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals undergoing liver transplantation due to end-stage liver disease caused by Hepatitis C Virus or alcoholic cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2008-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
serum FGL2 levels | various time points

CONTACTS AND LOCATIONS:
Overall Officials: Gary Levy, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital (University Health Network), Toronto, Ontario, Canada

REFERENCES:
- [Background] Shalev I, Liu H, Koscik C, Bartczak A, Javadi M, Wong KM, Maknojia A, He W, Liu MF, Diao J, Winter E, Manuel J, McCarthy D, Cattral M, Gommerman J, Clark DA, Phillips MJ, Gorczynski RR, Zhang L, Downey G, Grant D, Cybulsky MI, Levy G. Targeted deletion of fgl2 leads to impaired regulatory T cell activity and development of autoimmune glomerulonephritis. J Immunol. 2008 Jan 1;180(1):249-60. doi: 10.4049/jimmunol.180.1.249. PMID 18097026
- [Background] Liu H, Zhang L, Cybulsky M, Gorczynski R, Crookshank J, Manuel J, Grant D, Levy G. Identification of the receptor for FGL2 and implications for susceptibility to mouse hepatitis virus (MHV-3)-induced fulminant hepatitis. Adv Exp Med Biol. 2006;581:421-5. doi: 10.1007/978-0-387-33012-9_76. No abstract available. PMID 17037572
- [Background] Chan CW, Kay LS, Khadaroo RG, Chan MW, Lakatoo S, Young KJ, Zhang L, Gorczynski RM, Cattral M, Rotstein O, Levy GA. Soluble fibrinogen-like protein 2/fibroleukin exhibits immunosuppressive properties: suppressing T cell proliferation and inhibiting maturation of bone marrow-derived dendritic cells. J Immunol. 2003 Apr 15;170(8):4036-44. doi: 10.4049/jimmunol.170.8.4036. PMID 12682232